CLINICAL TRIAL: NCT00608335
Title: A Phase 1, Open-Label Study Of The Safety And Pharmacokinetics Of Repeated-Dose Micafungin (FK463) In Children (2-5 Years AND 6-11 Years) And Adolescents (12-16 Years) With Esophageal Candidiasis Or Other Invasive Candidiasis
Brief Title: Study of Mycamine® in Children With Fungal Infections to Evaluate Safety and Blood Levels of the Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9463-CL-2101
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Oropharyngeal Candidiasis; Candidemia; Invasive Candidiasis; Esophageal Candidiasis
Keywords: Antifungal; Micafungin; Echinocandin; Candidiasis
MeSH Terms: conditions — Candidemia; Candidiasis, Invasive; Candidiasis | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Micafungin 3.0 mg (Experimental): IV
  Interventions: Drug: Micafungin
- 2. Micafungin 4.5 mg (Experimental): IV
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: FK463

SUMMARY:
Children with fungal infections will be divided into two groups by weight. Children weighing < 25 kg will receive a higher dose of study medication (per kg body weight) for 10 to 14 days than children weighing > 25 kg.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, repeat-dose study conducted in two groups. Subjects in Group 1 and Group 2 will receive treatment for 10 to 14 days (per investigator clinical judgment); dose level (3.0 mg/kg or 4.5 mg/kg) will be determined by the subject's weight at baseline. Study procedures in both groups will be similar except that serial blood samples for assessment of pharmacokinetics will be collected in Group 1. Subjects may only participate in one group of the study.

At least 24 subjects, with at least 8 in each of three age ranges, will be enrolled in Group 1 (PK + safety). At least 36 subjects will be enrolled in Group 2 (safety), with at least 12 in each of the three age ranges.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 2 to 16 years inclusive
2. Subject has suspected, proven or probable candidiasis, candidemia or other invasive candidiasis
3. Subject has sufficient venous access to permit administration of study medication, collection of pharmacokinetic samples, and monitoring of laboratory safety variables

Exclusion Criteria:

1. Subject has evidence of significant liver disease, as defined by aspartate transaminase (AST), alanine transaminase (ALT), bilirubin or alkaline phosphatase > 5 times the upper limit of normal (ULN)
2. Subject has a concomitant medical condition that in the opinion of the investigator and/or medical monitor precludes enrollment into the study
3. Subject has a history of anaphylaxis, hypersensitivity, or any serious reaction to the echinocandin class of antifungals
4. Subject has received treatment with an echinocandin within one week prior to first dosing
5. Subject status is unstable and subject is unlikely to complete all study required procedures

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2007-10-14 (Actual); Primary Completion 2011-09-08 (Actual); Study Completion 2011-09-08 (Actual)

PRIMARY OUTCOMES:
PK parameters (AUCtau, Tmax, and Cmax) | 10 - 14 Days

SECONDARY OUTCOMES:
Adverse events | Day 1 to End of Study
Vital signs | Day 1 to End of Study
Hematology and chemistry laboratory tests | Day 1 to End of Study
12-lead ECGs and Physical examination | Day 1 to End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (13):
- United States (7):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Mercy Hospital, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- South Africa (6):
  - Benmed Park Clinic, Benoni
  - Grootte Schuur Hospital, Cape Town
  - GCT -Sunnyside Medi-clinic, Lynn East
  - St. Mary's Hospital, Mariannhill
  - Jubilee Hospital, Themba
  - 2 Military Hospital, Wynberg

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=260